CLINICAL TRIAL: NCT01601275
Title: Prospective Database of All Patients With Microbiologically Proven Mycobacteria Tuberculosis Infection Treated at Singapore General Hospital
Brief Title: Database of All Patients With Microbiologically Proven Mycobacteria Tuberculosis Infection
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/060/CTBdatabase
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Tuberculosis
Keywords: tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective data collection of all patients with microbiologically proven mycobacteria tuberculosis infection treated at Singapore General Hospital.

DETAILED DESCRIPTION:
Tuberculosis currently infects one third of the world's population and is responsible for killing approximately 2 million individuals annually. This is a major public health concern worldwide, and there has been a huge impetus to implement strategies for better tuberculosis control.

The investigators have established a system to track all patients with microbiologically proven tuberculosis treated at Singapore General Hospital, with vigilant recording and reporting systems, from the first instance when patients were diagnosed to the time they have completed anti-tuberculosis chemotherapy. The investigators endeavour to use this system to improve patient care by adopting patient-supportive approaches that lead to high compliance rates and best possible outcomes of treatment.

ELIGIBILITY:
Inclusion Criteria:

1) All patients with microbiologically proven mycobacteria tuberculosis infection treated at the Singapore General Hospital.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with microbiologically proven mycobacteria tuberculosis infection treated at the Singapore General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Actual)
Dates: Start 2012-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Final outcomes of patients who have been diagnosed with microbiologically proven mycobacteria tuberculosis infection at Singapore General Hospital | From diagnosis to final outcome

CONTACTS AND LOCATIONS:
Overall Officials: Su Ying Low, BMBCh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Dye C, Watt CJ, Bleed DM, Hosseini SM, Raviglione MC. Evolution of tuberculosis control and prospects for reducing tuberculosis incidence, prevalence, and deaths globally. JAMA. 2005 Jun 8;293(22):2767-75. doi: 10.1001/jama.293.22.2767. PMID 15941807
- [Background] DeAngelis CD, Flanagin A. Tuberculosis--a global problem requiring a global solution. JAMA. 2005 Jun 8;293(22):2793-4. doi: 10.1001/jama.293.22.2793. No abstract available. PMID 15941812